CLINICAL TRIAL: NCT05902299
Title: Modification of Antibiotic Susceptibility Testing: Evaluation of the Impact of This Change on Antibiotic Prescriptions at the Nancy Regional University Hospital
Brief Title: Evaluation of the Impact of the Modification of Antibiotic Susceptibility Testing on Antibiotic Prescriptions
Acronym: IPMRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CHARMILLON Alexandre, Ph.D., department of infectious and tropical diseases, Central Hospital, Nancy, France
Other Study IDs: 2022PI193
Record Dates: First submitted 2023-06-02; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Antibiotic Resistant Infection
Keywords: Antibiotic
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before antibiotic susceptibility testing
  Interventions: Drug: Antibiotic
- After antibiotic susceptibility testing

INTERVENTIONS:
Drug: Antibiotic — Evaluate the choice of antibiotic therapy prescribed for P. aeruginosa ou S. aureus infection
  Groups: Before antibiotic susceptibility testing

SUMMARY:
As of 2019, the CA-SFM (Comité de l'Antibiogramme de la Société Française de Microbiologie) recommends that the letter "I" or the term "intermediate" on antibiotic antibiograms. Instead, it is recommended that the term "sensible à forte posologie" or "SFP". These recommendations have been in place since 21/01/2022 at Nancy University Hospital.

Pseudomonas aeruginosa is the bacterium most affected by this change, as it has a high proportion of "high dosage" antibiotics.

Staphylococcus aureus is the most widely isolated bacterium, and also impacted by the change in antibiotic susceptibility testing.

The aim of this change in recommendations is to guarantee the efficacy of the proposed molecules.

Main objective Evaluate the impact of the change in antibiogram recommendations in samples positive for Pseudomonas aeruginosa and Staphylococcus aureus on antibiotic therapy (prescribed dosage)

Secondary objectives

* Evaluate the impact of changing the way antibiograms in Pseudomonas aeruginosa and Staphylococcus aureus on antibiotic therapy (molecule prescribed).
* Evaluate the impact of changing the way antibiograms on antibiotic therapy (molecule and dosage prescribed), depending on the strain identified (Pseudomonas aeruginosa or Staphylococcus aureus).
* Describe the impact of changing antibiograms in Pseudomonas aeruginosa and Staphylococcus aureus on antibiotic therapy (molecule and dosage prescribed) by department.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with a positive monobacterial P. aeruginosa or S.aureus resulting in an antibiotic susceptibility test between 01/03/2021 and 31/08/2021 (AVANT period) and between 01/03/2022 and 31/08/2022 (AFTER period)

Exclusion Criteria:

* patients from the maternity unit / the Centre Chirurgical Emile Gallé (CCEG) / dialysis department (UF 1094)
* patients with sample results that did not result in a prescription of antibiotics documented and duplicate samples relating to the same pathology and the same documented treatment
* patient opposed to research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients hospitalized who had a positive monobacterial sample for P. aeruginosa or S.aureus resulting in an antibiotic susceptibility test between 01/03/2021 and between 01/03/2021 and 31/08/2021 and between 01/03/2022 and 31/08/2022 and having received antibiotic therapy for this infection
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-07-03 (Estimated)

PRIMARY OUTCOMES:
comparison of dosage | Period before the introduction of the new antibiotic susceptibility test report (1 March to 31 August 2021) and after the introduction of the new antibiotic susceptibility test report (1 March to 31 August 2022)
  Dosage: number of DDDs (defined daily doses) / 1000 DH (hospitalization day). Dosage is calculated for all antibiotics, by class and then by molecule.

SECONDARY OUTCOMES:
comparison of prescription rates for antibiotics concerned | Period before the introduction of the new antibiotic susceptibility test report (1 March to 31 August 2021) and after the introduction of the new antibiotic susceptibility test report (1 March to 31 August 2022)
  Choice of molecule: antibiotic prescription rate of interest. The prescription rate will be calculated by class, then by molecule. Prescription rate = number of prescriptions of antibiotic X over the period / number of prescriptions of all antibiotics over the same period.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No